CLINICAL TRIAL: NCT00298935
Title: Pilot Clinical Trial of Osteopathic Manipulative Treatment (OMT) in Pregnancy
Brief Title: Study of the Effectiveness of Osteopathic Manipulative Treatment in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: Osteopathic Heritage Foundations (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-102
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Low Back Pain; Musculoskeletal Diseases; Pregnancy Complications
Keywords: Randomized Controlled Trial; Pregnant Women
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Diseases; Pregnancy Complications | interventions — Manipulation, Osteopathic

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment (OMT)

SUMMARY:
The purpose of this study is to determine whether osteopathic manipulative treatment (OMT):

* decreases pain and improves physical functioning in women during the third trimester of pregnancy
* decreases complications during obstetrical delivery
* improves quality of life in the post-partum period

DETAILED DESCRIPTION:
Women experience multiple changes in their anatomy and physiology during pregnancy that may cause pain and adversely affect quality of life. Additionally, about ten percent of women will experience signs and symptoms of pre-eclampsia or pre-term labor during their first pregnancy.

Preliminary studies of osteopathic manipulative treatment (OMT) have demonstrated a decrease in pain during pregnancy, although the mechanisms responsible for this effect are unclear.

Another theory is that osteopathic manipulative treatment (OMT) may help normalize sympathetic outflow, thereby minimizing pregnancy complications. A recently published retrospective study also suggests that pregnant women receiving osteopathic manipulative treatment (OMT) may be at lower risk for pre-term delivery and the presence of meconium during delivery.

ELIGIBILITY:
Inclusion Criteria:

* Third trimester pregnancy

Exclusion Criteria:

* High risk pregnancy
* Previous use of chiropractic manipulation, osteopathic manipulative treatment (OMT), physical therapy, or therapeutic ultrasound during the current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146
Dates: Start 2003-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for pain, Roland-Morris Disability Questionnaire, and SF-12 Health Status Survey during third trimester of pregnancy and continuing six weeks post-partum

SECONDARY OUTCOMES:
Occurrence of premature labor and delivery as well as obstetrical complications during delivery

CONTACTS AND LOCATIONS:
Overall Officials: John C. Licciardone, D.O., M.S., Principal Investigator — Osteopathic Research Center
Locations (1):
- Osteopathic Research Center, Fort Worth, Texas, United States